CLINICAL TRIAL: NCT01687257
Title: A Phase 2, Multicenter, Open-Label, Randomized Study to Investigate the Safety and Efficacy of GS-7977 and Ribavirin Administered for 48 Weeks in Patients Infected With Chronic HCV With Cirrhosis and Portal Hypertension With or Without Liver Decompensation
Brief Title: Sofosbuvir and Ribavirin in Patients With Chronic HCV With Cirrhosis and Portal Hypertension With or Without Liver Decompensation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0125; 2012-002457-29 (EudraCT Number)
Record Dates: First submitted 2012-09-12; First posted 2012-09-18 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C; Cirrhosis; Portal Hypertension; With or Without Liver Decompensation
MeSH Terms: conditions — Hepatitis C; Fibrosis; Hypertension, Portal | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF+RBV (Experimental): Participants will receive SOF+RBV for 48 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Observation, then SOF+RBV (Experimental): Participants will undergo 24 weeks of observation and then receive SOF+RBV for 48 additional weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — SOF 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study will evaluate the antiviral efficacy of combination therapy with sofosbuvir (SOF) plus ribavirin (RBV) for 48 weeks in adults with compensated and decompensated chronic hepatitis C virus (HCV) infection. Approximately 50 adults will be randomized (1:1) to receive study drug for 48 weeks or take part in an untreated observational arm for the first 24 weeks followed by study drug for another 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic infection with Hepatitis C with HCV RNA > 1000 IU/mL
* Individuals with cirrhosis with Child-Pugh score < 10
* Esophageal or gastric varices on endoscopy within 6 months prior to or at screening
* Hepatic Venous Pressure Gradient (HVPG) > 6 mmHg
* Body mass index (BMI) ≥ 18 kg/m^2
* Naïve to all nucleotides/nucleoside treatments for chronic HCV infection

Exclusion Criteria:

* Have any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance
* HIV or chronic hepatitis B virus (HBV) infection (HBsAg positive)
* Alpha-fetoprotein (AFP) > 50 unless negative imaging for hepatic masses within the last 6 months or during screening
* Refractory ascites as defined by requiring paracentesis > twice within 1 month prior to screening
* Active variceal bleeding within 6 months of screening
* Expected survival of < 1 year
* History of hepatorenal, or hepatopulmonary syndrome.
* Evidence of renal impairment (CrCl < 50 mL/min)
* History of major organ transplantation, including liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shampa De-Oertel, PhD, Study Director — Gilead Sciences
Locations (9):
- United States (4):
  - Aurora, Colorado
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Philadelphia, Pennsylvania
- Newtown, New South Wales, Australia
- Leclerc, Clichy, France
- Grafton, Auckland, New Zealand
- Spain (2):
  - Barcelona, Barcelona
  - Majadahonda, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Europe, Australia, and New Zealand. The first participant was screened on 27 November 2012. The last study visit occurred on 06 October 2015.
Pre-assignment Details: 63 participants were screened.
Groups:
- SOF+RBV (Group 1): Sofosbuvir (Sovaldi®; SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks
- Observation/SOF+RBV (Group 2; Not Treated): This reporting group only includes participants who were randomized to the Observation/SOF+RBV group who discontinued study prior to receiving study drug.
- Observation/SOF+RBV (Group 2; Received Treatment): This reporting group includes participants who completed observation and received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks.
Period: Overall Study
Arm/Group | SOF+RBV (Group 1) | Observation/SOF+RBV (Group 2; Not Treated) | Observation/SOF+RBV (Group 2; Received Treatment)
Started | 25 | 4 | 21
Completed | 17 | 0 | 15
Not Completed | 8 | 4 | 6
Not completed — Efficacy Failure | 6 | 0 | 5
Not completed — Subject Withdrew Consent | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Investigator's Discretion | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least 1 dose of study drug
Groups:
- SOF+RBV (Group 1): SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks
- SOF+RBV (Group 2; Received Treatment): This reporting group includes participants who completed observation and received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks.
- Total: Total of all reporting groups
Arm/Group | SOF+RBV (Group 1) | SOF+RBV (Group 2; Received Treatment) | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.2) | 56 (7.0) | 55 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 18 | 16 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 1 | 2
  White | 22 | 20 | 42
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for Region of Enrollment (n = 50).
  participants
    New Zealand | 2 | 4 | 6
    United States | 10 | 12 | 22
    France | 2 | 4 | 6
    Australia | 3 | 2 | 5
    Spain | 8 | 3 | 11
HCV Genotype [Number; unit: participants]
  Genotype 1a | 10 | 8 | 18
  Genotype 1b | 9 | 5 | 14
  Genotype 2a/2c | 1 | 0 | 1
  Genotype 2b | 1 | 1 | 2
  Genotype 3a | 2 | 6 | 8
  Genotype 4 | 1 | 1 | 2
  Genotype 4h | 1 | 0 | 1
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 3 | 6 | 9
    CT | 14 | 10 | 24
    TT | 8 | 5 | 13
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.1 (0.49) | 6.2 (0.79) | 6.1 (0.64)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 10 | 5 | 15
  ≥ 800,000 IU/mL | 15 | 16 | 31
Hepatic Venous Pressure Gradient (HVPG) [Mean (Standard Deviation); unit: mmHg] | 17.4 (4.70) | 16.4 (4.88) | 17.0 (4.85)
Child-Pugh-Turcotte (CPT) Score Category [Number; unit: participants] — CPT scores, widely used to grade the severity of cirrhosis and to determine the need for liver transplantation, are calculated based on a combination of laboratory values and clinical features. CPT scores can range from 5 to 15, with higher scores indicating a greater severity of disease.
  participants
    CPT A (5-6) | 8 | 10 | 18
    CPT B (7-10) | 17 | 11 | 28
Model for End-Stage Liver Disease (MELD) Score [Number; unit: participants] — MELD scores, used to assess prognosis and suitability for transplant, are calculated based on laboratory values only and can range from 6 to 40, with higher scores indicating greater disease severity.
  participants
    6 | 1 | 2 | 3
    7 | 0 | 3 | 3
    8 | 5 | 2 | 7
    9 | 3 | 1 | 4
    10 | 5 | 4 | 9
    11 | 0 | 4 | 4
    12 | 4 | 1 | 5
    13 | 2 | 1 | 3
    15 | 3 | 3 | 6
    16 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment. For the Observation/SOF+RBV group, SVR12 during the observational period was defined as HCV RNA < LLOQ for 12 consecutive weeks, any time during the observational period.
Time Frame: Posttreatment Week 12 (SOF+RBV) and up to 24 weeks (Observation)
Population: Participants who were randomized to the study.
Measure: Number; unit: percentage of participants
Groups:
- Observation Period (Group 2): 24 weeks of observation
- SOF+RBV (Group 2): Participants who completed observation and received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks
Arm/Group | SOF+RBV (Group 1) | Observation Period (Group 2) | SOF+RBV (Group 2)
Number analyzed (Participants) | 25 | 25 | 21
percentage of participants | 72.0 | 0 | 71.4

2. Secondary Outcome: Percentage of Participants With SVR at 4, 24, and 48 Weeks After Discontinuation of Therapy (SVR4, SVR24, and SVR48)
Description: SVR4, SVR24, and SVR48 were defined as HCV RNA < LLOQ at 4, 24, and 48 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4, 24, and 48
Population: Participants who were randomized and received at least 1 dose of study drug with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV (Group 1) | SOF+RBV (Group 2)
Number analyzed (Participants) | 25 | 21
percentage of participants
  SVR4 (Group 1: N = 25; Group 2: N = 21) | 72.0 | 76.2
  SVR24 (Group 1: N = 25; Group 2: N = 21) | 68.0 | 71.4
  SVR48 (Group 1: N = 17; Group 2: N = 13) | 94.1 | 100.0

3. Secondary Outcome: Percentage of Participants Experiencing On-Treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to 48 weeks
Population: Participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV (Group 1) | SOF+RBV (Group 2)
Number analyzed (Participants) | 25 | 21
percentage of participants | 8.0 | 0

4. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement.
Time Frame: Up to Posttreatment Week 24
Population: Participants who were randomized and received at least 1 dose of study drug with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV (Group 1) | SOF+RBV (Group 2)
Number analyzed (Participants) | 23 | 21
percentage of participants | 17.4 | 23.8

5. Secondary Outcome: Change From Baseline in Hepatic Venous Pressure Gradient (HVPG) at End of Treatment
Description: HVPG closely reflects the degree of portal hypertension in patients with cirrhosis. The end of treatment for the Observation group was defined as the end of the observation period. The treatment period for Group 2 was defined as the end of the observation period to the end of the treatment. Baseline values were the last available values on or prior to first dose date of any study drug.
Time Frame: Baseline; Week 24 (Observation) and Week 48 (SOF+RBV)
Population: Participants who were randomized to the study with available data at baseline and end of observation or end of treatment were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SOF+RBV (Group 1): SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for up to 48 weeks
- SOF+RBV (Group 2): SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for 48 weeks
- All SOF+RBV (Groups 1 and 2): Participants who received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 48 weeks in both Groups 1 and 2
Arm/Group | SOF+RBV (Group 1) | Observation Period (Group 2) | SOF+RBV (Group 2) | All SOF+RBV (Groups 1 and 2)
Number analyzed (Participants) | 19 | 21 | 18 | 37
mmHg | -1.6 (4.90) | 0.5 (2.52) | -0.4 (2.69) | -1.0 (3.97)

6. Secondary Outcome: Change From Baseline in Child-Pugh-Turcotte (CPT) Score
Description: CPT scores, widely used to grade the severity of cirrhosis and to determine the need for liver transplantation, are calculated based on a combination of laboratory values and clinical features. CPT scores can range from 5 to 15, with higher scores indicating a greater severity of disease. Data are presented as improvement, no change, or worsening in CPT scores at Week 24 (Observation) and Posttreatment Week 4 (SOF+RBV groups).
  Improvement in CPT score was defined as having a decrease in CPT score from baseline, no change in CPT score was defined as having no change in CPT score from baseline, and worsening in CPT score was defined as having an increase in CPT score from baseline.
  Baseline values were the last available values on or prior to first dose date of any study drug.
Time Frame: Baseline; Week 24 (Observation) and Posttreatment Week 4 (SOF+RBV)
Population: Participants who were randomized to the study with available data were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV (Group 2): SOF 400 mg tablet administered orally once daily + RBV tablets administered orally (1000 or 1200 mg daily based on weight) for up to 48 weeks
- All SOF+RBV (Groups 1 and 2): Participants who received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks in both Groups 1 and 2
Arm/Group | SOF+RBV (Group 1) | Observation Period (Group 2) | SOF+RBV (Group 2) | All SOF+RBV (Groups 1 and 2)
Number analyzed (Participants) | 23 | 20 | 18 | 41
percentage of participants
  Improvement in CPT Score | 65.2 | 10.0 | 38.9 | 53.7
  No Change in CPT Score | 26.1 | 75.0 | 50.0 | 36.6
  Worsening in CPT Score | 8.7 | 15.0 | 11.1 | 9.8

7. Secondary Outcome: Change From Baseline in Model for End Stage Liver Disease (MELD) Scores
Description: MELD scores, used to assess prognosis and suitability for transplant, are calculated based on laboratory values only and can range from 6 to 40, with higher scores indicating greater disease severity. Data are presented as improvement, no change, or worsening in MELD scores at Week 24 (Observation) and Posttreatment Week 4 (SOF+RBV groups).
  Improvement in MELD score was defined as having a baseline MELD score of 11-15 or 16-20 that changed to 0-10, or a baseline MELD score of 16-20 that changed to 11-15; no change in MELD score was defined as having no change in score group (0-10, 11-15, or 16-20) from baseline; and worsening in MELD score was defined as having a baseline MELD score of 0-10 that changed to 11-15 or 16-20, or a baseline MELD score of 11-15 that changed to 16-20.
  Baseline values were the last available values on or prior to first dose date of any study drug.
Time Frame: Baseline; Week 24 (Observation) and Posttreatment Week 4 (SOF+RBV)
Population: Participants who were randomized to the study with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV (Group 1) | Observation Period (Group 2) | SOF+RBV (Group 2) | All SOF+RBV (Groups 1 and 2)
Number analyzed (Participants) | 24 | 20 | 17 | 41
percentage of participants
  Improvement in MELD Score | 33.3 | 20.0 | 5.9 | 22.0
  No Change in MELD Score | 54.2 | 75.0 | 88.2 | 68.3
  Worsening in MELD Score | 12.5 | 5.0 | 5.9 | 9.8

ADVERSE EVENTS:
Time Frame: Up to 48 weeks plus 30 days
Description: Adverse event data includes all participants who were randomized to the study.
Groups:
- Observation Period Only (Group 2): This reporting group includes participants who were randomized to the Observation/SOF+RBV group and received up to 24 weeks of observation.
- SOF+RBV Treatment Only (Group 2): This reporting group includes participants who completed observation and received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for up to 48 weeks.
Arm/Group | SOF+RBV (Group 1) | Observation Period Only (Group 2) | SOF+RBV Treatment Only (Group 2)
Serious Adverse Events (participants affected / at risk) | 4/25 | 3/25 | 6/21
Other Adverse Events (participants affected / at risk) | 23/25 | 10/25 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (Group 1) (N=25) | Observation Period Only (Group 2) (N=25) | SOF+RBV Treatment Only (Group 2) (N=21)
Eye swelling (Eye disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (Group 1) (N=25) | Observation Period Only (Group 2) (N=25) | SOF+RBV Treatment Only (Group 2) (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 2
Ascites (Gastrointestinal disorders) | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 9 | 1 | 6
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Asthenia (General disorders) | 7 | 0 | 1
Fatigue (General disorders) | 6 | 1 | 9
Oedema peripheral (General disorders) | 0 | 3 | 5
Peripheral swelling (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 3
Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 7
Hepatic encephalopathy (Nervous system disorders) | 2 | 3 | 2
Memory impairment (Nervous system disorders) | 2 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 3
Insomnia (Psychiatric disorders) | 6 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years